CLINICAL TRIAL: NCT00549081
Title: DHEA Supplementation for Low Ovarian Response IVF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHEA for LR in IVF.CTIL
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Infertility, Female; In-Vitro Fertilization
Keywords: DHEA; IVF; low ovarian response
MeSH Terms: conditions — Infertility, Female | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IVF patients who had a low ovarian response in a previous hormonal-stimulation treatment, treated with recombinant FSH and LH.
  Interventions: Dietary Supplement: DHEA
- 2 (No Intervention): IVF patient who had a low ovarian response in a previous hormonal-stimulation treatment, treated with recombinant FSH and LH.

INTERVENTIONS:
Dietary Supplement: DHEA — oral DHEA tablets 75 mg daily
  Arms: 1

SUMMARY:
Approximately 10% of all couples will be diagnosed as infertile. The most efficient infertility treatment is In-Vitro Fertilization (IVF). One major determinant for success is production of an adequate number of oocytes (eggs) from the female in order to finally have good-quality embryos and finally acceptable pregnancy and delivery rates. Some women will not respond adequately to hormonal stimulation and will only a small number of oocytes. Therefore, the chances of finally having a successful delivery are significantly reduced. Although the specific definition of this situation is controversial, these patients are diagnosed as having "low ovarian response". This condition is more prevalent in older IVF patients as part of the reproductive aging process; it is possible at any age. Currently, the understanding of "low ovarian response" is limited, and although many therapeutic approaches have been suggested, no treatment has been proven significantly efficient.

DHEA is a pro-hormone produced by the adrenal gland and the ovary. DHEA serum levels become lower with age and in some chronic diseases. Therefore, some believe it may be beneficial as an 'anti-aging' factor. DHEA pills are available as a food-supplement, without need for prescription in the US.

DHEA is involved in the regulation of follicular growth in the ovaries. In a 2000 report, five IVF patients who had low ovarian response were treated with oral DHEA (Casson et al, Hum Reprod 2000;15:2129). A small increase in the ovarian response to hormonal stimulation was noticed. Barad and Gleicher reported their relatively extensive experience, summarizing treatment outcome in 25 IVF low-responders treated with oral DHEA pills (Barad and Gleicher, Hum Reprod 2006; 21, 2845). They observed increased increases in fertilized oocytes, normal day 3 embryos, and number of embryos transferred after DHEA treatment compared with a previous treatment outcome before DHEA.

Based on this observation, DHEA may appear useful for improving IVF outcome in some patients. However, a prospective randomized study on DHEA supplementation for IVF patients was not yet published. Our aim is to conduct such a study, focusing on IVF patient with low ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* IVF patient
* Low ovarian response to hormonal stimulation

Exclusion Criteria:

* Previous DHEA supplementation
* History of malignant disease
* Liver dysfunction
* Coagulation tendency

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2008-01; Study Completion 2008-12

PRIMARY OUTCOMES:
number of oocytes retrieved

SECONDARY OUTCOMES:
pregnancy rate delivery rate maximal serum estradiol levels ovarian reserve measures

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gonen, Principal Investigator — Meir Hospital, Sapir Medical Center, Kefar-Saba, Israel

REFERENCES:
- [Background] Barad D, Gleicher N. Effect of dehydroepiandrosterone on oocyte and embryo yields, embryo grade and cell number in IVF. Hum Reprod. 2006 Nov;21(11):2845-9. doi: 10.1093/humrep/del254. Epub 2006 Sep 22. PMID 16997936